CLINICAL TRIAL: NCT01837277
Title: Impact of a Dolutegravir-based Regimen on Early Mortality of Severely Immunocompromised AIDS Patients
Brief Title: Impact of a Dolutegravir-based Regimen on Early Mortality of AIDS Patients
Acronym: IDEA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fundação Bahiana de Infectologia (Other)
Responsible Party: Principal Investigator, Carlos Brites, Senior Investigator, Fundação Bahiana de Infectologia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SevereHIV
Record Dates: First submitted 2013-04-18; First posted 2013-04-23 (Estimated); Results first posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-03

CONDITIONS: Severely Immunocompromised HIV Patients
MeSH Terms: interventions — dolutegravir; efavirenz

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dolutegravir (Experimental): Intervention: Patients will receive ART regimen based on investigational drug Dolutegravir 50 mg QD + TDF 300 mg QD+ 3TC 150 mg BID
  Interventions: Drug: Dolutegravir 50 mg
- Efavirenz (Active Comparator): Intervention: Patients who received ART regimen based efavirenz (EFV 600 mg QD +TDF 300 mg QD+ 3TC 300 mg QD) for one year, befor the use of DTG as SOC for first-line therapy (historic controls)
  Interventions: Drug: Efavirenz-based regimens

INTERVENTIONS:
Drug: Dolutegravir 50 mg — Use of Dolutegravir -based regimens: patients will receive a Dolutegravir -based ART regimen (RAL 400 mg BID + TDF 300 mg QD + 3TC 150 mg BID)
  Other Names: Tivicay
  Arms: Dolutegravir
Drug: Efavirenz-based regimens — Efavirenz-based regimens: patients will receive an EFV-based regimen (EFV 600 mg QD + TDGF 300 mg QD + 3TC 300 mg QD)
  Other Names: Efavirenz
  Arms: Efavirenz

SUMMARY:
The current available antiretroviral (ARV) agents make possible a successful treatment of virtually all HIV-infected patients, but some problems related to early mortality are still of concern, mainly in resources-limited settings. There are several published reports showing that such patients are at a significantly higher risk of death during the first months of treatment, in comparison with the observed outcomes in developed countries. One of the consistently detected risks for early mortality across these reports is the baseline low CD4 count, although it does not seem to be the only reason for such outcome. In Brazil and other developing countries, there is still a large proportion of AIDS patients who are diagnosed with AIDS, or only seek health care for HIV infection late in the course of disease. Dolutegravir (DTG), the first HIV-1 integrase inhibitor, is a potent and safe ARV drug. The available evidence suggest it promotes a faster decline in HIV-1 plasma viremia, and a higher increase in CD4 cells count, in comparison with those in Efavirenz (EFV) arm. The investigators propose to compare the impact of DTG versus EFV in the early mortality rates for severely ill (CD4+ cells count <50 cells/mm3) patients starting ARV therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed HIV-1 infection (positive Western blot or plasma HIV-1 RNA >1,000 copies/ml)
* No previous use of any ARV drug (drug-naïve patients)
* Presence of clinical symptoms according to Rio de Janeiro / Caracas´ AIDS definition (Asthenia, Cachexia/Wasting, Cough, Dermatitis, persistent, Diarrhea, Fever, Lymphadenopathy, Candidiasis, oral, or hairy leukoplasia, Central nervous system dysfunction, Herpes zoster in individual younger than 60 years of age)), and/or any active AIDS-defining condition
* Baseline CD4+ cells count equal or lower than 50 cells/mm3
* Age equal or higher than 18 years
* HIV-1 plasma viral load ≥ 1,000 copies of HIV-1 RNA/ml

Exclusion Criteria:

* Undetectable plasma viral load at screening
* CD4 cells count>50 cells/mm3
* Asymptomatic individuals

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Brazil (3):
  - Fundação Bahiana de Infectologia/SEI, Salvador, Estado de Bahia
  - Universidade Federal do Rio de Janeiro, Rio de Janeiro, Rio de Janeiro
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dolutegravir | Efavirenz
Started | 92 | 92
Completed | 70 | 48
Not Completed | 22 | 44

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Efavirenz | Dolutegravir | Total
Number analyzed (Participants) | 92 | 92 | 184
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.3 (8.9) | 39.3 (11.5) | 38.3 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 63 | 96
  Male | 59 | 29 | 88
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 20 | 21 | 41
  Black | 15 | 5 | 20
  Asian | 1 | 0 | 1
  More than one race | 28 | 28 | 56
  Not reported | 28 | 48 | 76
Region of Enrollment [Count of Participants; unit: Participants]
  Brazil | 92 | 92 | 184
CD4 (cell/mm3) [Mean (Standard Deviation); unit: cells/mm3] | 23 (14) | 23 (14) | 23 (14)
Viral load (copies/mL [Median (Inter-Quartile Range); unit: log 10 copies/ml] | 5.6 [5.1 to 5.9] | 5.5 [5.0 to 5.9] | 5.5 [5.0 to 5.9]

OUTCOME MEASURES:

1. Primary Outcome: Early Mortality
Description: Proportion of deaths in each group
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Dolutegravir: Patients treated with Dolutegravir
- Efavirenz: Patients treated with Efavirenz
Arm/Group | Dolutegravir | Efavirenz
Number analyzed (Participants) | 92 | 92
Participants | 9 | 13

2. Secondary Outcome: Viral Load
Time Frame: 24 months
Reporting Status: Not Posted

3. Secondary Outcome: CD4 Count
Time Frame: 24 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events leading to interruption/change of ART in the 48 weeks period
Description: Proportion of adverse events leading to ART interruption were recorded, by group
Arm/Group | Dolutegravir | Efavirenz
All-Cause Mortality (participants affected / at risk) | 9/92 | 13/92
Serious Adverse Events (participants affected / at risk) | 9/92 | 13/92
Other Adverse Events (participants affected / at risk) | 0/92 | 11/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dolutegravir (N=92) | Efavirenz (N=92)
death (General disorders) | 9 | 13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dolutegravir (N=92) | Efavirenz (N=92)
CNS disturbances (Psychiatric disorders) | 0 | 11 — dizziness, sleep disturbance

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-01-06): https://cdn.clinicaltrials.gov/large-docs/77/NCT01837277/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-20): https://cdn.clinicaltrials.gov/large-docs/77/NCT01837277/SAP_001.pdf